CLINICAL TRIAL: NCT05662566
Title: Cohort Study: Risk of Failed Epidural in Patients With and Without Chronic Pain and Opioid Use Undergoing Laparotomy
Brief Title: Risk of Failed Epidural in Patients With and Without Chronic Pain and Opioid Use
Status: Completed | Type: Observational
Sponsor: Eske Kvanner Aasvang (Other)
Responsible Party: Sponsor-Investigator, Eske Kvanner Aasvang, Professor, MD, DMSci, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: WZ22042433
Record Dates: First submitted 2022-11-28; First posted 2022-12-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Postoperative Pain; Central Sensitisation
Keywords: Failed epidural; Chronic pain syndrome; Central Sensitization; Opioid use; Opioid Naive
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Chronic pain: Patients with chronic pain and fixed opioid use, undergoing laparotomy with epidural anesthesia as a part of the postoperative analgesic strategy
  Interventions: Procedure: Epidural replacement
- No chronic pain: Patients without chronic pain and without fixed opioid use, undergoing laparotomy with epidural anesthesia as a part of the postoperative analgesic strategy
  Interventions: Procedure: Epidural replacement

INTERVENTIONS:
Procedure: Epidural replacement — Insufficient analgesic effect of epidural anesthesia to the extent were replacement of the catheter is needed.
  Defined as insertion of a new epidural catheter

SUMMARY:
Patients with chronic pain syndrome (CPS) may develop central sensitization wich may lead to increased pain intensity and lower pain threshold sometimes to the extend of hyperalgesia and allodynia. Furthermore, patients with daily use of opioids may develop opioid tolerance, and to a lesser extent opioid induced hyperalgesia.

These factors may lead to a higher pain intensity in the perioperative setting resulting in the observed increased opioid dosage needed to treat the acute pain. Furthermore opioid titration may be difficult with higher levels of pain and a higher risk of opioid related adverse effects incl. respiratory depression and sedation.

The factors above advocate for utilizing opioid sparing analgesic techniques. In our department as in many others we use an multimodal opioid sparing approach for surgical procedures including epidural anesthesia (EA) as a standard part of the perioperative analgesia strategy after upper laparotomy, as a sufficient epidural anesthesia has shown to provide a stable and often better pain relief than systemic opioids in these patients.

Clinically, there is a suspicion that patients with CPS on fixed opioid treatment have a higher frequency of need for epidural optimization, despite the lack of an anatomical reason for this. One potential explanation could be an altered nociception, requesting another EA strategy than in non-opioid patients.

Purpose and hypothesis This study will explore the frequency of failed EA, defined as EA with insufficient analgesic effect to the extent were replacements of the epidural is needed within the first 5 postoperative days (PODs), testing the hypothesis that failed epidural occurs more frequent in patients with CPS on fixed opioid treatment than in non-opioid patients without CPS.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparotomy with epidural anesthesia as a part of the postoperative pain treatment
* For the intervention group - Patients with chronic pain disorder defined as pain for more than 3 months and a daily use of opioids regardless of dosage.
* For the control group - No chronic pain disorder defined as no daily use of opioid or other medicine with strong analgetic effect. A daily use of Acetaminophen and NSAIDs were deemed acceptable.

Exclusion Criteria:

* Patients with substance abuse
* Suspected withdrawal due to opioid deficiency - noted in the medical chart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with or without chronic pain and opioid use undergoing elective laparotomi with epidural anesthesia as a part of the postoperative pain treatment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Epidural replacement | 5 days postoperative
  Number of patients with the need of a new insertion of the epidural catheter

SECONDARY OUTCOMES:
Length of stay at the - post anaesthetic care unit (PACU) / Ward / Hospital | Total time of hospital stay up to 52 weeks
  Length of stay at post anaesthetic care unit / the surgical ward / entire admission. Defined from admission until discharged from the specific unit.
postoperative epidural optmisation | 5 days postoperative
  Return to the post anaesthetic care unit for epidural optimisation with medicine titration or retraction of the epidural catheter
Number of epidural replacements | 5 days postoperative
  Number of epidural replacements per patient

CONTACTS AND LOCATIONS:
Locations (1):
- Eske Kvanner Aasvang [eaasvang], Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No